CLINICAL TRIAL: NCT01571258
Title: Text4Diet: A Text Messaging Program for Weight Loss
Acronym: Text4Diet
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Santech, Inc (Industry)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Jennifer Shapiro, PhD, Scientific Director, Santech, Inc
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4R44CA138011 (NIH); 4R44CA138011 (NIH)
Record Dates: First submitted 2012-04-03; First posted 2012-04-05 (Estimated); Last update posted 2012-04-05 (Estimated); Status verified 2012-04

CONDITIONS: Text Messaging (Intervention); Control
Keywords: SMS; Obesity; Text Messaging; Intervention; Mobile Phone
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention)
- Text Messaging (Experimental): Participants in the intervention group will receive on average 4 texts per day consisting of weight related behavioral recommendations, knowledge based questions, and prompts to promote physical activity and weight monitoring. Texts are interactive and personally relevant based upon a baseline questionnaire.
  Interventions: Behavioral: Text Messaging

INTERVENTIONS:
Behavioral: Text Messaging — Participants in the intervention group will receive on average 4 texts per day consisting of weight related behavioral recommendations, knowledge based questions, and prompts to promote physical activity and weight monitoring. Texts are interactive and personally relevant based upon a baseline questionnaire.
  Arms: Text Messaging

SUMMARY:
The purpose of the present RCT is to evaluate a 12-month SMS intervention with expanded content, intervention strategies and interactive database logic, novel online enrollment, and automatic baseline scoring of measures to support a 12 month weight loss SMS intervention. The investigators hypothesized that the intervention group would have greater weight loss at 6 and 12 months than the control group and increased adherence to SMS would be associated with greater weight loss at 6 and 12 months.

DETAILED DESCRIPTION:
Background: Text messaging shows promise as an intervention mode for many health conditions due to its accessibility and timeliness . Few studies have evaluated the effectiveness of text message-based interventions for weight loss. This study is a randomized controlled trial comparing an intervention of daily text messaging (Text4Diet) focused on weight-related behaviors to a control group.

Participant Involvement: One hundred seventy overweight or obese adults will have their height and weight measured and complete a battery of questionnaires at baseline, 6 and 12 months. Participants in the intervention group will receive on average 4 texts per day consisting of weight related behavioral recommendations, knowledge based questions, and prompts to promote physical activity and weight monitoring. Texts are interactive and personally relevant based upon a baseline questionnaire. The control group will receive only monthly newsletters but not text messages. Participants in both conditions will receive monetary compensation for participation, travel to the study site, and reimbursements for text messaging.

Participants: Inclusion criteria consists of: a) age: 21 to 65 years, b) overweight or obese status: BMI between 25.0 and 39.9, c) regular access to the Internet, d) own and regularly use a cell phone and know how to use SMS, d) ability to read and speak English, and e) ability to participate in moderate PA. Exclusion criteria consists of a) current pregnancy or the intention of becoming pregnant during the 12 month trial, b) moving out of the country during the 12 month trial, and c) current eating disorder.

Dates: Recruitment for the RCT began in September 2010. The RCT began in January 2011 and ended in December 2011. Data analysis will occur through June 2012.

Location: San Diego, CA

Risks to Participants: This study involves low risk. Participation may involve some discomforts, such as embarrassment from sharing information about home environment, weight, and technology, diet, and exercise habits. There is a risk of loss of confidentiality of research information. All risks will be minimized according to the study protocol.

ELIGIBILITY:
Inclusion Criteria:

* age: 21 to 65 years
* overweight or obese status: BMI between 25.0 and 39.9
* regular access to the Internet
* own and regularly use a cell phone and know how to use SMS
* ability to read and speak English
* ability to participate in moderate PA.

Exclusion Criteria:

* current pregnancy or the intention of becoming pregnant during the 12 month trial
* moving out of the country during the 12 month trial
* current eating disorder

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2010-09; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Weight | 6 months, 12 months
  We will assess the difference in weight loss between the intervention and the control group at 6 months and 12 months.

SECONDARY OUTCOMES:
Pedometer Steps/Day | 6 months, 12 months
  Change in average pedometer steps per day in the intervention group.
Adherence | 6 months, 12 months
  Level of adherence in responding to SMS. We also will investigate the correlation between adherence and weight loss.
Treatment Satisfaction | 6 months and 12 months
  We will assess satisfaction with the SMS intervention in the intervention group only.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Shapiro, PhD, Study Director — Santech, Inc
Locations (1):
- Santech, Inc., San Diego, California, United States